CLINICAL TRIAL: NCT04567758
Title: The Effect of Telerehabilitation on Clinical Results, Patient Expectation, Motivation and Satisfaction Level in Patients With Chronic Low Back Pain
Brief Title: The Effect of Telerehabilitation in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Fatih ÖZDEN, Principal Investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2020.518
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-02

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Telerehabilitation; Pain; Quality of Life; Motivation; Expectation; Patient Satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants, outcomes assessor, and the analyzer of the statistics of the study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (TR) Group (Experimental): The TR group will be followed up through the video-based exercise software within the 8-week home exercise program.
  Interventions: Other: Telerehabilitation
- Conventional Rehabilitation (CR) Group (Active Comparator): The CR group will be trained face-to-face with conventional methods before the 8-week home exercise program, and an exercise program will be prescribed with a visual information form.
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The home exercise program includes the following exercises:
  1. Lumbar region and lower extremity stretching exercises;
  2. Exercises to strengthen the abdominal muscles;
  3. Exercises to strengthen the lumbar muscles;
  4. Bridging, spine mobility exercise, McKenzie extension, and Williams flexion exercises
  A web-based telerehabilitation platform (Fizyoweb) will be used to deliver the exercise program. Using the Fizyoweb web application, exercises will be presented to the patients in the form of audio-video and detailed instructions with explanations. The exercise program to be given will be prescribed specifically with slight changes according to the patient's condition. The exercise protocol will be the same as in the conventional rehabilitation group. Patients will be asked to do the exercises once a day for 8 weeks and 10 repetitions each.
  Other Names: TR
  Arms: Telerehabilitation (TR) Group
Other: Conventional Rehabilitation — The home exercise program, which will be given with conventional rehabilitation, will be educated to the patient in the clinic on the first day. Exercise information form including explanation and picture of the exercises will be given to the patients. The exercise program to be given will be prescribed specifically with slight changes according to the patient's condition. Patients will be asked to do the exercises once a day for 8 weeks and 10 repetitions each.
  The home exercise program includes the following exercises:
  1. Lumbar region and lower extremity stretching exercises;
  2. Exercises to strengthen the abdominal muscles;
  3. Exercises to strengthen the lumbar muscles;
  4. Bridging, spine mobility exercise, McKenzie extension, and Williams flexion exercises
  Other Names: CR
  Arms: Conventional Rehabilitation (CR) Group

SUMMARY:
Telerehabilitation enables patients to easily adapt to home exercise programs and to be monitored remotely by their clinicians. The aim of this study is to investigate the effectiveness of the home exercise program, which is integrated into 8-week remote asynchronous video telerehabilitation sessions, on clinical status in terms of pain, functionality, quality of life parameters, as well as patient expectation, motivation, and satisfaction levels.

DETAILED DESCRIPTION:
Low back pain is symptomatic pathology in the region between the twelve ribs and lower gluteal line defined as the lumbar region and sometimes accompanied by radicular symptoms spreading to the lower extremity, but it is not considered as a pathology alone. They are evaluated and treated on the basis of symptom duration, potential cause, the presence or absence of radicular symptoms, and the corresponding anatomical or radiographic abnormalities. Exercise is considered an essential element in the management of physical therapy and rehabilitation in patients with chronic low back pain. However, it has been found in the studies that improvements after physical therapy and rehabilitation applications are not preserved in the long term, and recurrence of chronic low back pain is common. In order to prevent this, physiotherapists need to follow their patients for a long time and to participate in the rehabilitation process. With a more cost-effective treatment model such as telerehabilitation, patients can be followed up more efficiently during home exercise. The aim of this study is to investigate the effectiveness of the home exercise program, which is integrated into 8-week remote asynchronous video telerehabilitation sessions, on clinical status in terms of pain, functionality, quality of life parameters, as well as patient expectation, motivation, and satisfaction levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65
* Patients who have complained of low back pain for at least 3 months
* Pain and numbness that does not spread to the legs

Exclusion Criteria:

* Patients with cognitive disorders or communications problems to complete assessments or treatment interventions.
* Individuals who have undergone surgical operations on the spine and/or extremities
* Specific pathological conditions (e.g. malignancy, fracture, systemic rheumatoid disease)
* Orthopedic and neurological problems that prevent evaluation and/or treatment
* Complaints of pain and numbness spreading to the lower extremities
* Individuals with a diagnosed psychiatric illness
* Individuals who have received physiotherapy in the last 6 months
* Individuals who use another treatment method during the study
* Individuals with musculoskeletal pain in any other part of the body during work
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 minutes
  Visual Analogue Scale (VAS): The patients will be asked to mark their pain feelings for rest and activity on a 10 cm numerical line (0: no pain, 10: unbearable pain). It is planned to use numerical VAS in our study. The cut-off values for chronic musculoskeletal pain will be classified as the severity of pain according to VAS as follows:
  <3.4 centimeters: mild pain, 3.5-7.4 centimeters: moderate pain, > 7.5 centimeters: severe pain.
Five Repeated Sit-to-Stand Test | 5 minutes
  In the starting position, the participant will be asked to sit in a chair without a standard armrest, with his back flat, feet shoulder-width apart and soles flat on the floor, with his arms crossed in front of the chest. With the "start" command, the participant is asked to stand up straight from the chair and return to the starting position without disturbing the arm position. Up to 5 repetitions are recorded in seconds.
Timed Up and Go Test | 5 minutes
  The patient stands up from a sitting position, walks on a 3-meter line, turns back and sits on the chair again. The duration of the performance is recorded in seconds.
Oswestry Disability Index (ODI) | 5 minutes
  ODI is a questionnaire consisting of 10 questions measuring the functional status. Each question is evaluated between 0-5 points and the total maximum score is 50. As the total score increases, functionality decreases and disability increases.
Tampa Kinesiophobia Scale (TSK) | 5 minutes
  TSK is a questionnaire consisting of 17 questions and used in the evaluation of kinesiophobia (fear of movement). 4-point Likert scale (1 = Strongly disagree, 4 = Strongly agree) is used. The scale is scored between 17-68. The high score the person gets on the scale indicates that his kinesiophobia is also high.
Short Form-36 (SF-36) | 5 minutes
  SF-36 consists of thirty-six items. These provide measurements of eight dimensions. Subscales evaluate health between 0-100 points; '0' indicates poor health, '100' indicates good health.
System Usability Scale (SUS) | 5 minutes
  SUS is an evaluation tool developed to evaluate systems or software in terms of usability, expectation, and satisfaction. The SUS, which is a 5-point Likert-type scale, includes 10 items in total. At the end of the scale, a score between 0 and 100 is obtained.

SECONDARY OUTCOMES:
Exercise Adherence Rating Scale (EARS) | 5 MİNUTES
  EARS provides a measurement of commitment to home exercise. This may facilitate the evaluation of interventions that promote self-management, for the treatment of chronic conditions.
Exercise Diary | 2 minutes
  The patients will be asked to fill the daily exercise diary chart, whether the they have done the exercise or not in order to follow up their home exercise program.
Expectation and satisfaction assessment | 5 minutes
  The expectation questionnaire will be conducted on the day of the start of the home exercise program, and the satisfaction questionnaire will be carried out on the day of termination from the two questionnaires prepared by the researchers of the study for the assessment of expectations and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Zübeyir Sarı, PT, PhD, Study Chair — Marmara University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Kötekli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No